CLINICAL TRIAL: NCT00251823
Title: The Safety and Efficacy of Eptifibatide-Facilitated Percutaneous Coronary Angioplasty Versus Primary Percutaneous Coronary Angioplasty Alone
Brief Title: Safety and Efficacy Study of Eptifibatide in Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Schering-Plough (Industry); Medtronic (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO4319
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Myocardial Infarction
Keywords: ST-Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

INTERVENTIONS:
Drug: Eptifibatide facilitated PCI

SUMMARY:
Rationale:

ST-elevation myocardial infarction (STEMI) is usually triggered by rupture of an atherosclerotic plaque that then accumulates platelets and fibrin and leads to an occlusive coronary thrombus. Clinical benefits obtained with revascularization of the infarct related artery (IRA) depend on the achievement of four goals:

1. Early reperfusion
2. Full restoration of normal flow in the epicardial vessels
3. Full restoration of flow in the microcirculation, and
4. Preservation of myocardial function.

Reperfusion of the IRA can be achieved pharmacologically with intravenous thrombolytic agents, or mechanically with percutaneous coronary intervention (PCI). In Canada, thrombolysis is the current standard of care in most hospitals, although there is mounting evidence that primary PCI is superior, and many Canadian centres are shifting towards this strategy. To offer primary PCI to community hospitals without on site cardiac catheterization facilities, regional programs need to be present that allow rapid transfer to invasive centers that offer this procedure round-the-clock.

Recent evidence suggests that angiographic and clinical results with primary PCI could be further enhanced by facilitation with a pharmacological treatment given prior to the procedure. The present proposal plans to examine the safety and efficacy of eptifibatide to facilitate coronary angioplasty in STEMI in patients who present to centres with and without on-site catheterization facilities.

The primary outcome measure will be a composite clinical endpoint including death, recurrent myocardial infarction, recurrent unstable ischemia, or stroke, at 30 days.

Secondary endpoints include the percent thrombolysis in myocardial infarction (TIMI) grade 3 coronary flow after the PCI, myocardial perfusion score, individual clinical outcomes as listed for the primary endpoint, resolution of ST-segment elevation, requirement for subsequent revascularization, frequency of congestive heart failure (CHF), cardiogenic shock, and Canadian Cardiovascular Society (CCS) angina class.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic chest discomfort of 30 minutes duration
* Onset of chest pain 12 hours prior to entry into the study
* ST segment elevation of > 1 mm (0.1 mV) in two or more contiguous electrocardiographic leads (on a standard 12 lead electrocardiogram [ECG]), or left bundle branch block not known to be old

Exclusion Criteria:

* Active bleeding
* History of stroke within 90 days or any intracranial bleed.
* Major surgery or trauma within the past 6 weeks
* Uncontrolled hypertension (systolic blood pressure [SBP] 200 mm Hg and/or diastolic blood pressure [DBP] 110 mm Hg despite treatment)
* Prolonged (> 10 minutes) cardiopulmonary resuscitation
* Inadequate vascular access
* PCI within the last 30 days
* Thrombolytic agents within the preceding 7 days
* Concurrent use of warfarin
* A blood coagulation disorder (i.e. international normalized ratio [INR] > 2.0, platelet count < 100,000/mm3, or hematocrit < 30%)
* Intolerance to aspirin or clopidogrel
* A subcutaneous therapeutic dose of any low molecular weight heparin (LMWH) within 12 hours
* Known severe contrast allergy
* Other medical condition that is likely to result in death within 12 months
* Participation in a study or another investigational device or drug trial within the past four weeks
* Pregnancy
* Known severe renal impairment (creatinine > 200 mole/l)
* Sustained hypotension, systolic blood pressure < 80 mm Hg, or the need for intravenous (IV) inotropes and/or intraaortic balloon counterpulsation to support the blood pressure
* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-07; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary clinical endpoint is a composite measure of clinical outcomes of death, recurrent myocardial infarction, and recurrent severe ischemia, which will be assessed at 30 days after the index acute myocardial infarction (AMI)

SECONDARY OUTCOMES:
Determine if a facilitated PCI strategy with early initiation of eptifibatide improves the percentage of patients with TIMI grade 3 flow measured at the time of baseline angiography
improves post procedural TIMI perfusion scoreC
improves ST-segment elevation resolution, a surrogate marker of clinical efficacy
improves left ventricular (LV) ejection fraction
improves functional capacity
decreases subsequent revascularization (PCI , or coronary artery bypass graft [CABG])

CONTACTS AND LOCATIONS:
Overall Officials: Michel R. Le May, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Zeymer U, Zahn R, Schiele R, Jansen W, Girth E, Gitt A, Seidl K, Schroder R, Schneider S, Senges J. Early eptifibatide improves TIMI 3 patency before primary percutaneous coronary intervention for acute ST elevation myocardial infarction: results of the randomized integrilin in acute myocardial infarction (INTAMI) pilot trial. Eur Heart J. 2005 Oct;26(19):1971-7. doi: 10.1093/eurheartj/ehi293. Epub 2005 Apr 27. PMID 15857851